CLINICAL TRIAL: NCT05935878
Title: Cemented Versus Cementless Unicompartmental Knee Arthroplasty (UKA) - A Single-blind Randomised Controlled Trial
Brief Title: Cemented Versus Cementless Unicompartmental Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, David W Murray, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID7088
Record Dates: First submitted 2023-06-08; First posted 2023-07-07 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee Arthroplasty; Unicompartmental; Fixation; Radiostereometric Analysis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to receive either a cementless or cemented Oxford Unicompartmental Knee Arthroplasty.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Cementless Oxford Unicompartmental Knee Arthroplasty (Experimental): Phase III Cementless Oxford Unicompartmental Knee Replacement (Biomet)
  Interventions: Device: Cementless Oxford Unicompartmental Knee Arthroplasty
- Cemented Oxford Unicompartmental Knee Arthroplasty (Active Comparator): Phase III Cemented Oxford Unicompartmental Knee Replacement (Biomet)
  Interventions: Device: Cemented Oxford Unicompartmental Knee Arthroplasty

INTERVENTIONS:
Device: Cementless Oxford Unicompartmental Knee Arthroplasty — All patients will undergo the same surgical approach. 0.8mm diameter tantalum marker balls will be placed in the tibia and femur in all cases. Cementless components have a hydroxy-appatite coating to facilitate bone ingrowth. The cementless femoral component also has a smaller second peg, located anteriorly to the larger central peg that is also present of the cemented femoral component.
  Other Names: Cementless Oxford Unicompartmental Knee Replacement
  Arms: Cementless Oxford Unicompartmental Knee Arthroplasty
Device: Cemented Oxford Unicompartmental Knee Arthroplasty — All patients will undergo the same surgical approach. 0.8mm diameter tantalum marker balls will be placed in the tibia and femur in all cases. All cemented components will be secured using the same cement.
  Other Names: Cemented Oxford Unicompartmental Knee Replacement
  Arms: Cemented Oxford Unicompartmental Knee Arthroplasty

SUMMARY:
Unicompartmental knee replacement for selected cases of osteoarthritis is less invasive than total knee replacement. It gives better range of movement; patients stay for shorter time in the hospital and have a more natural feel than total knee replacement. Usually, the implant is fixed in the bone using bone cement. However, there are potential disadvantages of using bone cement. The operation takes longer; cement can get squeezed out into the surrounding tissues and may interfere with function. To avoid these problems, the implant can be fixed without cement. Cementless components have a special coating to encourage bone in-growth and fixation. Although the investigators believe cementless fixation will be at least as good as cemented fixation, there is a risk that it could be worse and might result in loosening.

The aim of this study is therefore to compare the outcome of cemented and cementless unicompartmental knee replacement.

DETAILED DESCRIPTION:
Design: A prospective, randomised trial to compare the outcome of cemented and cementless unicompartmental knee replacement.

Size: 40 subjects in total will be recruited with 20 in each arm.

Methods: Patients will be recruited from the routine waiting list for unicompartmental knee replacement at the Nuffield Orthopaedic Centre. All subjects will have the procedure explained and be fully consented prior to the procedure.

Randomisation: Patients will be randomly allocated to receive either a cemented or cementless Oxford Unicompartmental Knee Replacement. This will be performed using a randomisation program based on optimisation (Minim). Subjects will be stratified according to sex and age.

Operation: All subjects will undergo the same surgical approach. 0.8mm Tantalum marker balls will be placed at standardised sites on the femur and tibia in all cases. All cemented components will be secured using the same cement. Cementless components have a hydroxy-appatite coating to facilitate bone ingrowth.

Follow-up: All patients will be followed up at 0, 3, 6, 12, 24, 60, and 120 months with clinical and radiological assessment. Clinical assessment will involve documentation with the Oxford Knee Score. Patients will undergo radiostereometric analysis and fluoroscopy to study implant migration and occurence of radiolucency, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects with osteoarthritis of knee fulfilling the standard indications for an Oxford Unicompartmental Knee Replacement.
* American Society of Anaesthesiologists (ASA) Score of 1 to 3.

Exclusion Criteria:

* Subjects with severe limiting systemic illness (i.e. ASA > 3).
* Subjects who are too large for radiostereometric analysis to be carried out.
* Subjects who have had previous open surgery or anterior cruciate ligament (ACL) reconstruction on the same knee.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2002-11-08 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Murray, MA, MD, FRCS, Principal Investigator — University of Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kendrick BJ, Kaptein BL, Valstar ER, Gill HS, Jackson WF, Dodd CA, Price AJ, Murray DW. Cemented versus cementless Oxford unicompartmental knee arthroplasty using radiostereometric analysis: a randomised controlled trial. Bone Joint J. 2015 Feb;97-B(2):185-91. doi: 10.1302/0301-620X.97B2.34331. PMID 25628280
- [Result] Campi S, Kendrick BJL, Kaptein BL, Valstar ER, Jackson WFM, Dodd CAF, Price AJ, Murray DW. Five-year results of a randomised controlled trial comparing cemented and cementless Oxford unicompartmental knee replacement using radiostereometric analysis. Knee. 2021 Jan;28:383-390. doi: 10.1016/j.knee.2020.09.003. Epub 2021 Jan 4. PMID 33408039
- See also: Publication of 2-year results — https://boneandjoint.org.uk/article/10.1302/0301-620X.97B2.34331
- See also: Abstract of the (partial) 10-year results — https://boneandjoint.org.uk/Article/10.1302/1358-992X.2022.7.086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A consecutive series of patients awairing an Oxford Unicompartmental Knee Replacement (OUKR) were invited to participate in the study. Consenting participants received an OUKR between November 2008 and March 2010 at the Nuffield Orthopaedic Centre (Oxford, UK).
Period: Overall Study
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Started | 23 | 24
1 Year | 22 | 21
2 Years | 22 | 21
5 Years | 19 | 20
10 Years | 16 | 15
Completed | 16 | 15
Not Completed | 7 | 9
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Revision of implant | 1 | 1
Not completed — Mobile bearing dislocation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 15 | 13 | 28
Age, Continuous [Mean (Full Range); unit: years] | 67.7 [49.1 to 81.6] | 65.9 [49.5 to 79.5] | 66.7 [49.1 to 81.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 14 | 12 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Radiostereometric Analysis Examination - Translations
Description: Patients will have weight-bearing stereoradiographs. These stereoradiographs will be analysed using model-based radiostereometric analysis which will allow the migration of the components relative to the bone to be determined. Three-dimensional translations will be measured in millimetres. The component position at the post-operative timepoint was used as the baseline for measurement of migration. Migration can be interpreted as:
  * X translation: Positive (+ve) = Medial; Negative (-ve) = Lateral
  * Y translation: Positive (+ve) = Superior; Negative (-ve) = Inferior
  * Z translation: Positive (+ve) = Anterior; Negative (-ve) = Posterior
Time Frame: Patients will be examined 3 months post surgery.
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
millimetres
  Femoral X Migration | -0.01 (0.36) | 0.05 (0.40)
  Femoral Y Migration | -0.10 (0.34) | -0.17 (0.25)
  Femoral Z Migration | 0.26 (0.48) | 0.14 (0.33)
  Tibial X Migration | -0.09 (0.22) | 0.08 (0.28)
  Tibial Y Migration | -0.23 (0.18) | -0.10 (0.17)
  Tibial Z Migration | -0.03 (0.20) | -0.02 (0.26)

2. Primary Outcome: Radiostereometric Analysis Examination - Translations
Description: as for outcome 1
Time Frame: Patients will be examined 6 months post surgery.
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
millimetres
  Femoral X Migration | -0.12 (0.31) | 0.05 (0.28)
  Femoral Y Migration | -0.02 (0.39) | -0.02 (0.39)
  Femoral Z Migration | 0.24 (0.39) | 0.16 (0.29)
  Tibial X Migration | 0.06 (0.19) | 0.06 (0.19)
  Tibial Y Migration | -0.28 (0.17) | 0.06 (0.18)
  Tibial Z Migration | -0.03 (0.13) | -0.05 (0.30)

3. Primary Outcome: Radiostereometric Analysis Examination - Translations
Description: as for outcome 1
Time Frame: Patients will be examined 12 months post surgery.
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
millimetres
  Femoral X Translation | -0.18 (0.28) | 0.05 (0.28)
  Femoral Y Translation | -0.12 (0.24) | -0.12 (0.25)
  Femoral Z Translation | 0.26 (0.31) | 0.24 (0.32)
  Tibial X Translation | -0.04 (0.21) | 0.01 (0.24)
  Tibial Y Translation | -0.28 (0.19) | -0.09 (0.19)
  Tibial Z Translation | -0.01 (0.15) | 0.00 (0.26)

4. Primary Outcome: Radiostereometric Analysis Examination - Translations
Description: as for outcome 1
Time Frame: Patients will be examined 24 months post surgery.
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
millimetres
  Femoral X Translation | -0.05 (0.53) | 0.03 (0.34)
  Femoral Y Translation | -0.04 (0.27) | -0.05 (0.32)
  Femoral Z Translation | 0.21 (0.23) | 0.22 (0.42)
  Tibial X Translation | 0.01 (0.19) | 0.06 (0.26)
  Tibial Y Translation | -0.34 (0.23) | -0.13 (0.23)
  Tibial Z Translation | -0.02 (0.16) | 0.03 (0.22)

5. Primary Outcome: Radiostereometric Analysis Examination - Translations
Description: Patients will have weight-bearing stereoradiographs. These stereoradiographs will be analysed using model-based radiostereometric analysis which will allow the migration of the components relative to the bone to be determined. Three-dimensional translations will be measured in millimetres.
Time Frame: Patients will be examined 60 months post surgery.
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 19 | 20
millimetres
  Femoral X Translation | -0.02 (0.46) | 0.10 (0.35)
  Femoral Y Translation | -0.07 (0.29) | -0.16 (0.19)
  Femoral Z Translation | 0.14 (0.31) | 0.20 (0.30)
  Tibial X Translation | -0.03 (0.21) | 0.03 (0.22)
  Tibial Y Translation | -0.28 (0.19) | -0.14 (0.29)
  Tibial Z Translation | 0.00 (0.11) | 0.01 (0.31)

6. Primary Outcome: Radiostereometric Analysis Examination - Translations
Description: as for outcome 1
Time Frame: Patients will be examined 120 months post surgery.
Population: 1 Cemented Oxford Unicompartmental Knee Arthroplasty could not be analysed due poor quality stereoradiographs with obstruction of bone markers being obstructed. Consequently, although 15 Cemented Oxford Unicompartmental Knee Arthroplasties were followed-up at 120 months, only 14 could be analysed.
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 16 | 14
millimetres
  Femoral X Translation | -0.12 (0.50) | 0.24 (0.31)
  Femoral Y Translation | -0.14 (0.27) | -0.16 (0.21)
  Femoral Z Translation | 0.20 (0.36) | 0.14 (0.28)
  Tibial X Translation | 0.00 (0.26) | 0.00 (0.16)
  Tibial Y Translation | -0.29 (0.20) | -0.15 (0.42)
  Tibial Z Translation | -0.01 (0.21) | 0.02 (0.23)

7. Primary Outcome: Radiostereometric Analysis Examination - Rotations
Description: Patients will have weight-bearing stereoradiographs. These stereoradiographs will be analysed using model-based radiostereometric analysis which will allow the migration of the components relative to the bone to be determined. Three-dimensional rotations will be measured in degrees.The component position at the post-operative timepoint was used as the baseline for measurement of migration. Migration can be interpreted as:
  *For the Femoral Component* X Rotation: Positive (+ve) = Increased Flexion; Negative (-ve) = Decreased Flexion Y Rotation: Positive (+ve) = Internal Rotation; Negative (-ve) = External Rotation Z Rotation: Positive (+ve) = Valgus; Negative (-ve) = Varus
  *For the Tibial Component* X Rotation: Positive (+ve) = Reduced Slope; Negative (-ve) = Increased Slope Y Rotation: Positive (+ve) = Internal Rotation; Negative (-ve) = External Rotation Z Rotation: Positive (+ve) = Valgus; Negative (-ve) = Varus
Time Frame: Patients will be examined at 3 months post surgery.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
Degrees
  Femoral X Rotation | 0.22 (0.95) | 0.19 (0.47)
  Femoral Y Rotation | 0.26 (0.55) | 0.10 (0.74)
  Femoral Z Rotation | -0.16 (0.89) | -0.10 (0.95)
  Tibial X Rotation | -0.48 (0.88) | -0.09 (0.50)
  Tibial Y Rotation | 0.05 (0.63) | -0.08 (0.46)
  Tibial Z Rotation | 0.36 (0.70) | -0.10 (0.68)

8. Primary Outcome: Radiostereometric Analysis Examination - Rotations
Description: Patients will have weight-bearing stereoradiographs. These stereoradiographs will be analysed using model-based radiostereometric analysis which will allow the migration of the components relative to the bone to be determined. Three-dimensional rotations will be measured in degrees.The component position at the post-operative timepoint was used as the baseline for measurement of migration. Migration can be interpreted as:
  * For the Femoral Component* X Rotation: Positive (+ve) = Increased Flexion; Negative (-ve) = Decreased Flexion Y Rotation: Positive (+ve) = Internal Rotation; Negative (-ve) = External Rotation Z Rotation: Positive (+ve) = Valgus; Negative (-ve) = Varus
  * For the Tibial Component* X Rotation: Positive (+ve) = Reduced Slope; Negative (-ve) = Increased Slope Y Rotation: Positive (+ve) = Internal Rotation; Negative (-ve) = External Rotation Z Rotation: Positive (+ve) = Valgus; Negative (-ve) = Varus
Time Frame: Patients will be examined at 6 months post surgery.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
Degrees
  Femoral X Rotation | 0.04 (0.56) | 0.27 (0.81)
  Femoral Y Rotation | 0.48 (0.79) | 0.05 (0.62)
  Femoral Z Rotation | -0.11 (0.90) | 0.19 (0.76)
  Tibial X Rotation | -0.46 (0.78) | -0.25 (0.65)
  Tibial Y Rotation | 0.12 (0.58) | 0.07 (0.36)
  Tibial Z Rotation | 0.33 (0.71) | 0.15 (0.98)

9. Primary Outcome: Radiostereometric Analysis Examination - Rotations
Description: as for outcome 8
Time Frame: Patients will be examined at 12 months post surgery.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
Degrees
  Femoral X Rotation | 0.22 (0.57) | 0.16 (0.65)
  Femoral Y Rotation | 0.24 (0.52) | -0.05 (0.63)
  Femoral Z Rotation | -0.26 (0.93) | 0.25 (0.80)
  Tibial X Rotation | -0.38 (0.73) | -0.10 (0.70)
  Tibial Y Rotation | 0.16 (0.54) | -0.02 (0.45)
  Tibial Z Rotation | 0.10 (0.63) | -0.29 (0.67)

10. Primary Outcome: Radiostereometric Analysis Examination - Rotations
Description: as for outcome 8
Time Frame: Patients will be examined at 24 months post surgery.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
Degrees
  Femoral X Migration | 0.20 (0.54) | 0.23 (0.68)
  Femoral Y Migration | 0.23 (0.52) | 0.32 (0.52)
  Femoral Z Migration | 0.00 (1.28) | -0.06 (0.75)
  Tibial X Migration | -0.40 (0.76) | -0.17 (0.69)
  Tibial Y Migration | 0.24 (0.61) | 0.03 (0.44)
  Tibial Z Migration | -0.01 (0.60) | -0.31 (0.68)

11. Primary Outcome: Radiostereometric Analysis Examination - Rotations
Description: as for outcome 8
Time Frame: Patients will be examined at 60 months post surgery.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 19 | 20
Degrees
  Femoral X Rotation | 0.35 (0.44) | 0.16 (0.54)
  Femoral Y Rotation | 0.29 (0.79) | -0.34 (2.07)
  Femoral Z Rotation | -0.17 (1.14) | 0.25 (0.88)
  Tibial X Rotation | -0.28 (0.80) | -0.34 (1.19)
  Tibial Y Rotation | 0.28 (0.47) | 0.07 (0.40)
  Tibial Z Rotation | -0.13 (0.68) | -0.45 (0.80)

12. Primary Outcome: Radiostereometric Analysis Examination - Rotations
Description: as for outcome 8
Time Frame: Patients will be examined at 120 months post surgery.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 16 | 14
Degrees
  Femoral X Rotation | -0.02 (0.50) | 0.27 (0.55)
  Femoral Y Rotation | 0.19 (0.79) | 0.38 (0.81)
  Femoral Z Rotation | 0.53 (0.90) | 0.38 (1.16)
  Tibial X Rotation | -0.43 (0.74) | -0.66 (2.59)
  Tibial Y Rotation | 0.18 (0.48) | 0.15 (0.36)
  Tibial Z Rotation | -0.50 (0.64) | -0.79 (1.14)

13. Primary Outcome: Radiostereometric Analysis Examination - Maximum Total Point Motion
Description: Patients will have weight-bearing stereoradiographs. These stereoradiographs will be analysed using model-based radiostereometric analysis which will allow the migration of the components relative to the bone to be determined. Maximum Total Point Motion (MTPM - defined as the length of the translation vector of the point of the component model that has migrated the most) will be measured in millimetres.
Time Frame: Patients will be examined at 3 months post surgery.
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
millimetres
  Femoral MTPM | 0.93 (0.67) | 0.80 (0.36)
  Tibial MTPM | 0.84 (0.45) | 0.61 (0.40)

14. Primary Outcome: Radiostereometric Analysis Examination - Maximum Total Point Motion
Description: as for outcome 13
Time Frame: Patients will be examined at 12 months post surgery.
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
millimetres
  Femoral MTPM | 0.76 (0.35) | 0.80 (0.53)
  Tibial MTPM | 0.78 (0.37) | 0.65 (0.45)

15. Primary Outcome: Radiostereometric Analysis Examination - Maximum Total Point Motion
Description: as for outcome 13
Time Frame: Patients will be examined at 24 months post surgery.
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
millimetres
  Femoral MTPM | 0.87 (0.42) | 0.94 (0.87)
  Tibial MTPM | 0.84 (0.39) | 0.64 (0.51)

16. Primary Outcome: Radiostereometric Analysis Examination - Maximum Total Point Motion
Description: as for outcome 13
Time Frame: Patients will be examined at 60 months post surgery.
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 19 | 20
millimetres
  Femoral MTPM | 0.87 (0.40) | 0.95 (0.88)
  Tibial MTPM | 0.79 (0.30) | 0.80 (0.68)

17. Primary Outcome: Radiostereometric Analysis Examination - Maximum Total Point Motion
Description: as for outcome 13
Time Frame: Patients will be examined at 120 months post surgery.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 16 | 14
millimetres
  Femoral MTPM | 0.98 (0.41) | 0.84 (0.41)
  Tibial MTPM | 0.82 (0.32) | 0.95 (1.33)

18. Primary Outcome: Radiographic Examination
Description: Fluoroscopic imaging will be used to study the occurence of radiolucencies beneath the components. Anteroposterior radiographs will be analysed to assess the presence and position of radiolucencies. Radiolucencies will be graded as either 'no radiolucency present', 'partial radiolucency', or 'complete radiolucency'.
Time Frame: Patients will be examined at 12 months post surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
Participants
  Tibial Component: Partial Radiolucency | 7 | 11
  Tibial Component: Complete Radiolucency | 1 | 2
  Tibial Component: No Radiolucency | 14 | 8
  Femoral Component: Partial Radiolucency | 0 | 0
  Femoral Component: Complete Radiolucency | 0 | 0
  Femoral Component: No Radiolucency | 22 | 21

19. Primary Outcome: Radiographic Examination
Description: as for outcome 18
Time Frame: Patients will be examined at 24 months post surgery.
Population: Plain radiographs were only available for 21 of the 22 Cementless Oxford Unicompartmental Knee Arthroplasties at the 60 month timepoint, which explains the discrepency between the number of patients analyzed and the number of patients reported in the patient flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 21 | 21
Participants
  Tibial Component: Partial Radiolucency | 6 | 8
  Tibial Component: Complate Radiolucency | 0 | 5
  Tibial Component: No Radiolucency | 15 | 8
  Femoral Component: Partial Radiolucency | 0 | 0
  Femoral Component: Complate Radiolucency | 0 | 0
  Femoral Component: No Radiolucency | 21 | 21

20. Primary Outcome: Radiographic Examination
Description: as for outcome 18
Time Frame: Patients will be examined at 60 months post surgery.
Population: Plain radiographs were only available for 18 of the 20 Cemented Oxford Unicompartmental Knee Arthroplasties at the 60 month timepoint, which explains the discrepency between the number of patients analyzed and the number of patients reported in the patient flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 19 | 18
Participants
  Tibial Component: Partial Radiolucency | 1 | 6
  Tibial Component: Complete Radiolucency | 0 | 1
  Tibial Component: No Radiolucency | 18 | 11
  Femoral Component: Partial Radiolucency | 0 | 0
  Femoral Component: Complete Radiolucency | 0 | 0
  Femoral Component: No Radiolucency | 19 | 18

21. Primary Outcome: Radiographic Examination
Description: as for outcome 18
Time Frame: Patients will be examined at 120 months post surgery.
Population: Plain radiographs were only available for 15 of the 16 Cementless Oxford Unicompartmental Knee Arthroplasties and 14 of the 15 Cemented Oxford Unicompartmental Knee Arthroplastiesat the 60 month timepoint, which explains the discrepency between the number of patients analyzed and the number of patients reported in the patient flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 15 | 14
Participants
  Tibial Component: Partial Radiolucency | 1 | 6
  Tibial Component: Complete Radiolucency | 0 | 0
  Tibial Component: No Radiolucency | 14 | 8
  Femoral Component: Partial Radiolucency | 0 | 0
  Femoral Component: Complete Radiolucency | 0 | 0
  Femoral Component: No Radiolucency | 15 | 14

22. Primary Outcome: Clinical Assessment
Description: Clinical assessment will involve documentation with the Oxford Knee Score. The score will be calculated on a scale of 0 (worst) to 48 (best).
Time Frame: Patients will be assessed pre-operatively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 23 | 24
score on a scale | 24 (7) | 23 (6)

23. Primary Outcome: Clinical Assessment
Description: as for outcome 22
Time Frame: Patients will be assessed at 12 months post surgery.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
score on a scale | 41 [28 to 48] | 40 [20 to 47]

24. Primary Outcome: Clinical Assessment
Description: as for outcome 22
Time Frame: Patients will be assessed at 24 months post surgery.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
score on a scale | 42 [24 to 48] | 38 [20 to 47]

25. Primary Outcome: Clinical Assessment
Description: as for outcome 22
Time Frame: Patients will be assessed at 60 months post surgery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 20 | 19
score on a scale | 41 (7) | 37 (12)

26. Primary Outcome: Clinical Assessment
Description: as for outcome 22
Time Frame: Patients will be assessed at 120 months post surgery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 16 | 14
score on a scale | 42 (7) | 39 (10)

27. Primary Outcome: Radiostereometric Analysis Examination - Maximum Total Point Motion
Description: as for outcome 13
Time Frame: Patients will be assessed at 6 months post surgery.
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
Number analyzed (Participants) | 22 | 21
millimetres
  Femoral MTPM | 0.86 (0.43) | 0.80 (0.44)
  Tibial MTPM | 0.79 (0.42) | 0.64 (0.45)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected out to 10 years follow-up.
Arm/Group | Cementless Oxford Unicompartmental Knee Arthroplasty | Cemented Oxford Unicompartmental Knee Arthroplasty
All-Cause Mortality (participants affected / at risk) | 1/23 | 2/24
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/24
Other Adverse Events (participants affected / at risk) | 0/23 | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cementless Oxford Unicompartmental Knee Arthroplasty (N=23) | Cemented Oxford Unicompartmental Knee Arthroplasty (N=24)
Implant Revision (Surgical and medical procedures) | 1 (1) | 1 (1) — Revision surgery involving the replacement of one or more of the implant components.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cementless Oxford Unicompartmental Knee Arthroplasty (N=23) | Cemented Oxford Unicompartmental Knee Arthroplasty (N=24)
Mobile Bearing Dislocation (Surgical and medical procedures) | 0 (0) | 1 (1) — Dislocation of the mobile bearing which normally articulates with the femoral and tibial components of the Oxford Unicompartmental Knee Replacement.

LIMITATIONS AND CAVEATS:
At 10 years, loss to follow-up meant there were less than 16 knees in each group required by the power calculation for the study.

Maximum Total Point Motion (MTPM) was used as an overall indicator of migration, however the utility of MTPM is limited as it compounds measurement errors so tends to overestimate migration.

As the study was powered to detect differences in migration using RSA, the patient numbers were too small to detect differences in clinical outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2009-09-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT05935878/Prot_SAP_000.pdf
  • Informed Consent Form (2002-05-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT05935878/ICF_001.pdf